CLINICAL TRIAL: NCT04322838
Title: Tromsø Birch Rust Allergy Study. Allergy to Birch Rust Fungi, a Possible Explanation to Seasonal Airway Allergy During Autumn? A Pilot Study With 30 Patients With Suspected Allergy to Birch Rust and 15 Non-allergic Controls.
Brief Title: Tromsø Birch Rust Allergy Study. Allergy to Birch Rust, a Possible Explanation to Seasonal Airway Allergy During Autumn?
Acronym: Tro-BRA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of North Norway (Other)
Collaborators: Luxembourg Institute of Health (Other Government); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sørensen, Department leader, University Hospital of North Norway
Other Study IDs: 62924 (REK)
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hypersensitivity, Immediate; Allergy
Keywords: Birch rust fungi; Melampsoridium Betulinum; Allergy; Allergic rhino-conjunctivitis; Allergic asthma
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity | interventions — Patch Tests; Nasal Provocation Tests; Basophil Degranulation Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for measurement of specific IgE Full blood for Basophil Activation Test (BAT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 30 patients with self-reported seasonal allergic airway symptoms in the period from 1st of August to 15.th of october
  Interventions: Diagnostic Test: MeDALL questionnaire for allergic diseases; Diagnostic Test: Registration of allergic symptoms; Diagnostic Test: Skin Prick Test; Diagnostic Test: Specific IgE in serum; Diagnostic Test: Nasal provocation test; Diagnostic Test: Basophil Activation Test
- Controls: 15 non-allergic individuals
  Interventions: Diagnostic Test: MeDALL questionnaire for allergic diseases; Diagnostic Test: Registration of allergic symptoms; Diagnostic Test: Skin Prick Test; Diagnostic Test: Specific IgE in serum; Diagnostic Test: Nasal provocation test; Diagnostic Test: Basophil Activation Test

INTERVENTIONS:
Diagnostic Test: MeDALL questionnaire for allergic diseases — Questionnaire about allergic symptoms and disease
  Other Names: Mechanisms of the development of allergy
Diagnostic Test: Registration of allergic symptoms — Daily registration of allergic symptoms from eyes, nose and lungs on scale from 0-10 and daily registration of use of anti allergic medication from 1st of August to 15th of October.
Diagnostic Test: Skin Prick Test — Diagnostic skin test for sensitization to allergens
Diagnostic Test: Specific IgE in serum — Diagnostic test for sensitization to allergens in serum
  Other Names: IgE
Diagnostic Test: Nasal provocation test — Diagnostic test for allergic rhinitis. Patients and controls are exposed to an allergen with a nasal spray. Allergic reactions are measured with Linder score and Pean Nasal Inspiratory Flow (PNIF)
Diagnostic Test: Basophil Activation Test — Basophil leukocytes are extracted from full blood and exposed to 6 different doses of allergen and activation of basophils are measured.
  Other Names: BAT

SUMMARY:
In this project we study if spores from birch rust fungi (Melampsoridium Betulinum = MB) may be the eliciting allergen in patients with seasonal airway allergy during autumn in North Norway. Patients with suspected allergy to MB are compared with non-allergic controls using data about allergic disease and daily allergic symptoms during autumn. Daily spread of MB spores are compared with daily variations in allergic symptoms. Sensitization to MB and MB allergy are tested with skin prick test, specific immunoglobulin E (IgE) in serum, nasal provocation test and basophil activation test (BAT).

DETAILED DESCRIPTION:
It is unknown why patients experience seasonal airway allergy during autumn in Norway, when there is no spread of pollen. Some old studies indicate that rust fungi on other plants may act as allergens to humans (1-6). In Norway, some patients report typical symptoms of allergic rhino-conjunctivitis and asthma from August to October which stops when temperature falls below zero (Celsius). Based on several patient experiences we hypothesize that MB may cause seasonal airway allergy during autumn. In this pilot study we will compare 30 patients with suspected allergy to MB with a control group of 15 non-allergic individuals. All 45 participants will answer the MeDALL (mechanisms of the development of allergy) questionnaire (7) about allergic diseases and daily register allergic symptoms (8) in the period from 1st of August to 15th of October 2020. Daily variations in symptoms will be compared with daily variations in spread of MB spores registered in pollen traps. Sensitization to MB will be tested with skin prick test and specific IgE in serum and allergy to MB with nasal provocation test and basophil activation test (BAT).

Identification of allergens and production of MB extracts for testing will be performed by Luxembourg institute of Health (LiH)(9-12) and BAT by Oslo University hospital (13-14)

ELIGIBILITY:
Inclusion Criteria:

* Self reported seasonal airway allergic symptoms during autumn

Exclusion Criteria:

* Perennial airway allergic symptoms without worsening during autumn

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with allergic symptoms of allergic rhino-conjunctivitis and/or allergic asthma in the period from 1st of august to 15th of October.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Allergy to Birch rust fungi | 1st of August to 15th of October 2020
  Allergic symptoms during spread of Birch rust spores and positive sensitization and nasal provocation test to birch rust fungi.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sørensen, PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Cadham,F.T., Asthma due to grain rusts. Jama, 1924, 83(1):p.27.
- [Background] Waldbott, G.L.A., M.S., Rust and Smut, Major causes of respiratory allergy. Ann Intern Med., 1940. 14(2):p.215-224
- [Background] Croce MA, da Costa Manso ER, Gambale W, Takayama L, Oliveira Andrade CE, Pereira Pinto JH, Morato Castro FF, Croce J. Sensitization to the fungus Hemileia vastatrix (coffee leaf rust). Allergy. 2001 Jul;56(7):684-7. doi: 10.1034/j.1398-9995.2001.00053.x. PMID 11421929
- [Background] Simon-Nobbe B, Denk U, Poll V, Rid R, Breitenbach M. The spectrum of fungal allergy. Int Arch Allergy Immunol. 2008;145(1):58-86. doi: 10.1159/000107578. Epub 2007 Aug 20. PMID 17709917
- [Background] Horner WE, Lopez M, Salvaggio JE, Lehrer SB. Basidiomycete allergy: identification and characterization of an important allergen from Calvatia cyathiformis. Int Arch Allergy Appl Immunol. 1991;94(1-4):359-61. doi: 10.1159/000235403. PMID 1937899
- [Background] Gupta, D.A., Environmental and occupational respiratory diseases - 1033. Rust fungi of plants and high IgE levels in asymptomatic workers of a stored food grains godown: a possible relationship. World Allergy Organization Journal, 2013. 6(suppl 1):p.32.
- [Background] Hohmann C, Pinart M, Tischer C, Gehring U, Heinrich J, Kull I, Melen E, Smit HA, Torrent M, Wijga AH, Wickman M, Bachert C, Lodrup Carlsen KC, Carlsen KH, Bindslev-Jensen C, Eller E, Esplugues A, Fantini MP, Annesi-Maesano I, Momas I, Porta D, Vassilaki M, Waiblinger D, Sunyer J, Anto JM, Bousquet J, Keil T; MeDALL Study Group. The development of the MeDALL Core Questionnaires for a harmonized follow-up assessment of eleven European birth cohorts on asthma and allergies. Int Arch Allergy Immunol. 2014;163(3):215-24. doi: 10.1159/000357732. Epub 2014 Mar 1. PMID 24642608
- [Background] Bousquet J, Devillier P, Anto JM, Bewick M, Haahtela T, Arnavielhe S, Bedbrook A, Murray R, van Eerd M, Fonseca JA, Morais Almeida M, Todo Bom A, Menditto E, Passalacqua G, Stellato C, Triggiani M, Ventura MT, Vezzani G, Annesi-Maesano I, Bourret R, Bosse I, Caimmi D, Cartier C, Demoly P, Just J, Portejoie F, Siroux V, Viart F, Bergmann KC, Keil T, Klimek L, Mosges R, Pfaar O, Shamai S, Zuberbier T, Mullol J, Valero A, Spranger O, Tomazic PV, Kowalski ML, Kuna P, Kupczyk M, Raciborski F, Samolinski B, Toppila-Salmi SK, Valovirta E, Cruz AA, Sarquis-Serpa F, da Silva J, Stelmach R, Larenas-Linnemann D, Rodriguez Gonzalez M, Burguete Cabanas MT, Kvedariene V, Valiulis A, Chavannes NH, Fokkens WJ, Ryan D, Sheikh A, Bachert C, Hellings PW, VandenPlas O, Ballardini N, Kull I, Melen E, Westman M, Wickman M, Bindslev-Jensen C, Eller E, Bosnic-Anticevich S, O'Hehir RE, Agache I, Bieber T, Casale T, Gemicioglu B, Ivancevich JC, De Vries G, Sorensen M, Yorgancioglu A, Laune D; MACVIA working group. Daily allergic multimorbidity in rhinitis using mobile technology: A novel concept of the MASK study. Allergy. 2018 Aug;73(8):1622-1631. doi: 10.1111/all.13448. Epub 2018 Apr 24. PMID 29569295
- [Background] Sorensen M, Kuehn A, Mills ENC, Costello CA, Ollert M, Smabrekke L, Primicerio R, Wickman M, Klingenberg C. Cross-reactivity in fish allergy: A double-blind, placebo-controlled food-challenge trial. J Allergy Clin Immunol. 2017 Oct;140(4):1170-1172. doi: 10.1016/j.jaci.2017.03.043. Epub 2017 May 4. No abstract available. PMID 28479332
- [Background] Schiener M, Hilger C, Eberlein B, Pascal M, Kuehn A, Revets D, Planchon S, Pietsch G, Serrano P, Moreno-Aguilar C, de la Roca F, Biedermann T, Darsow U, Schmidt-Weber CB, Ollert M, Blank S. The high molecular weight dipeptidyl peptidase IV Pol d 3 is a major allergen of Polistes dominula venom. Sci Rep. 2018 Jan 22;8(1):1318. doi: 10.1038/s41598-018-19666-7. PMID 29358620
- [Background] Kuehn A, Codreanu-Morel F, Lehners-Weber C, Doyen V, Gomez-Andre SA, Bienvenu F, Fischer J, Ballardini N, van Hage M, Perotin JM, Silcret-Grieu S, Chabane H, Hentges F, Ollert M, Hilger C, Morisset M. Cross-reactivity to fish and chicken meat - a new clinical syndrome. Allergy. 2016 Dec;71(12):1772-1781. doi: 10.1111/all.12968. Epub 2016 Jul 15. PMID 27344988
- [Background] Kuehn A, Hilger C, Lehners-Weber C, Codreanu-Morel F, Morisset M, Metz-Favre C, Pauli G, de Blay F, Revets D, Muller CP, Vogel L, Vieths S, Hentges F. Identification of enolases and aldolases as important fish allergens in cod, salmon and tuna: component resolved diagnosis using parvalbumin and the new allergens. Clin Exp Allergy. 2013 Jul;43(7):811-22. doi: 10.1111/cea.12117. PMID 23786287
- [Background] Dahlen B, Nopp A, Johansson SG, Eduards M, Skedinger M, Adedoyin J. Basophil allergen threshold sensitivity, CD-sens, is a measure of allergen sensitivity in asthma. Clin Exp Allergy. 2011 Aug;41(8):1091-7. doi: 10.1111/j.1365-2222.2011.03763.x. Epub 2011 Apr 25. PMID 21518044
- [Background] Hoffmann HJ, Santos AF, Mayorga C, Nopp A, Eberlein B, Ferrer M, Rouzaire P, Ebo DG, Sabato V, Sanz ML, Pecaric-Petkovic T, Patil SU, Hausmann OV, Shreffler WG, Korosec P, Knol EF. The clinical utility of basophil activation testing in diagnosis and monitoring of allergic disease. Allergy. 2015 Nov;70(11):1393-405. doi: 10.1111/all.12698. Epub 2015 Sep 8. PMID 26198455